CLINICAL TRIAL: NCT03978221
Title: Diaphragm Performance Evaluation With Tissue Doppler Ultrasound Examination During Spontaneous Breathing in Facial Mask and During Non-invasive Ventilation in the Post-extubation Period.
Brief Title: Tissue Doppler Ultrasound During Spontaneous Breathing and Non-invasive Ventilation in the Post-extubation Period.
Acronym: TDIpostext
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Gianmaria Cammarota, Principal Investigator, MD of ICU staff, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 22/19
Record Dates: First submitted 2019-05-13; First posted 2019-06-07 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-05

CONDITIONS: Acute Respiratory Failure; Non-invasive Ventilation
Keywords: Diaphragmatic Tissue Doppler; Non invasive ventilation; Spontaneous breathing; Post-extubation

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diaphragmatic tissue doppler evaluation (Experimental): A tissue Doppler evaluation, using a sectorial probe, will be performed by analyzing the diaphragmatic displacement velocity during inspiration and expiration randomly assessed in spontaneous breathing with Venturi Mask and in Non-invasive ventilation with a helmet or facial mask
  Interventions: Other: Post-extubation TDI

INTERVENTIONS:
Other: Post-extubation TDI — A diaphragmatic tissue Doppler evaluation will be performed during non-invasive ventilation and spontaneous breathing trial applied in random sequence. Each trial will last 20 minutes. During the last minute of each trial a tissue doppler diaphragmatic examination will be performed to assess the speed of diaphragmatic displacement during inspiration and expiration.

SUMMARY:
The aim of the present investigation will be to evaluate diaphragmatic excursion velocity during non-invasive ventilation and spontaneous breathing at both inspiration and expiration.

this analysis will be performed through diaphragmatic tissue Doppler assessment.

DETAILED DESCRIPTION:
Early weaning from invasive ventilation, in patients admitted to intensive care, is associated with a marked reduction in ventilator-associated pneumonia, length of stay in intensive care unit and hospital, total duration of mechanical ventilation and decrease in overall mortality. Moreover, in case of need of protected extubation, non-invasive ventilation has allowed to prevent re-intubation and decrease hospital mortality compared to the simple administration of oxygen through a facial mask, in particular when applied immediately after extubation.

The diaphragmatic tissue doppler imaging (TDI) is an ultrasonographic technique derived from ultrasound evaluation of the heart's motility. It can be easily used on the diaphragm to calculate the speed of muscles displacement that could be associated with patient's respiratory drive.

The aim of the study is the evaluation of the diaphragmatic excursion velocity variations using diaphragmatic tissue doppler, measured in venturi mask and non-invasive ventilation in the post-extubation period, in order to compare the diaphragm stress variations during the two different modes.

Method Patients after extubation will be randomly submitted to a spontaneous breathing test in venturi mask and in facemask or helmet NIV.

Each trial will last 20 minutes. During the last minute of each trial a tissue doppler diaphragm examination will be performed to assess the speed speed of muscle displacement, acceleration and deceleration.

Inclusion criteria: invasive mechanical ventilation > 24h with consequent extubation.

Exclusion criteria: refusal to grant consent, pregnancy, age < 18 years, haemodynamic instability, difficult management of secretions, required inotropic and / or vasoactive drugs at high doses.

During the study, vital parameters will be given.

ELIGIBILITY:
Inclusion Criteria:

* invasive mechanical ventilation > 24h with consequent extubation

Exclusion Criteria:

* refusal to grant consent
* pregnancy
* age >18 years
* haemodynamic instability
* difficult management of secretions
* required inotropic and / or vasoactive drugs at high doses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-12 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
diaphragmatic displacement velocity | through each trial completion, an average of 20 minutes
  Inspiratory and expiratory diaphragmatic displacement velocity evaluated with tissue doppler during the NIV trial and in spontaneous breathing with Venturi mask.

SECONDARY OUTCOMES:
Diaphragmatic acceleration | through each trial completion, an average of 20 minutes
  Inspiratory and expiratory diaphragmatic displacement acceleration evaluated with tissue doppler during the NIV trial and in spontaneous breathing with Venturi mask.
Gas exchange - arterial carbon dioxide tension | through each trial completion, an average of 20 minutes
  PaCO2, will be obtained performing ABG sample
Gas exchange - pH | through each trial completion, an average of 20 minutes
  pH will be obtained performing ABGs.
Gas exchange - arterial oxygen tension | through each trial completion, an average of 20 minutes
  arterial oxygenation PaO2 will be obtained performing ABGs.
Dyspnea level | through each trial completion, an average of 20 minutes
  dyspnea level evaluated through visual analogical scale ( VAS dyspnea)
Comfort level | through each trial completion, an average of 20 minutes
  Comfort level evaluated through Comfort Scale
Hemodynamic parameters, Heart Rate (HR) | athrough each trial completion, an average of 20 minutes
  Heart Rate (HR)
Blood Pressure (BP) | through each trial completion, an average of 20 minutes
  invasive Mean arterial Blood Pressure

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U Maggiore della Carità, Novara, Italy

REFERENCES:
- [Background] Vaschetto R, Longhini F, Persona P, Ori C, Stefani G, Liu S, Yi Y, Lu W, Yu T, Luo X, Tang R, Li M, Li J, Cammarota G, Bruni A, Garofalo E, Jin Z, Yan J, Zheng R, Yin J, Guido S, Della Corte F, Fontana T, Gregoretti C, Cortegiani A, Giarratano A, Montagnini C, Cavuto S, Qiu H, Navalesi P. Early extubation followed by immediate noninvasive ventilation vs. standard extubation in hypoxemic patients: a randomized clinical trial. Intensive Care Med. 2019 Jan;45(1):62-71. doi: 10.1007/s00134-018-5478-0. Epub 2018 Dec 10. PMID 30535516